CLINICAL TRIAL: NCT05384691
Title: A Phase II, Open-label, Single Arm Study to Evaluate the Efficacy of Luspatercept in Erythropoiesis-stimulating Agent Naive Lower-risk MDS Patients With or Without Ring Sideroblasts Who do Not Require RBC Transfusions
Brief Title: Efficacy of Luspatercept in ESA-naive LR-MDS Patients With or Without Ring Sideroblasts Who do Not Require Transfusions
Acronym: LENNON
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Anne Sophie Kubasch, Coordinating Investigator, University of Leipzig
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LENNON Trial
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Myelodysplastic Syndromes; Anemia
Keywords: MDS; Anemia; Ring sideroblast; Low risk; non-transfusion dependence (NTD)
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia | interventions — luspatercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Luspatercept (Other): Single-arm design: All patients are treated with 1.75 mg Luspatercept per kg body weight subcutaneously on day 1 of each 21 day cycle for up to 24 weeks and in case of response for up to 1.5 years.
  Interventions: Drug: Luspatercept Injection

INTERVENTIONS:
Drug: Luspatercept Injection — All formally included patients will receive 1.75 mg/kg luspatercept administered subcutaneously every three weeks (on day 1 of each 21-day cycle) for a duration of 24 weeks.
  Responders at the response assessment (according to HI-E) in week 25 will be further treated with 1.75 mg/kg luspatercept until loss of response for an expected maximum of 18 months.
  Other Names: LUS

SUMMARY:
Anemia in patients with very low, low or intermediate risk myelodysplastic syndromes (MDS), that are non-transfusion dependent

DETAILED DESCRIPTION:
Patients with very low, low or intermediate risk myelodysplastic syndromes (MDS) presenting with anemia, transfusion independence (NTD) and naive towards ESA treatment

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of myelodysplastic syndrome (MDS) according to WHO classification
* Very low-, low-, or intermediate-risk disease MDS with up to 3.5 according to revised International Prognostic Scoring System (IPSS-R)
* Less than 5% blasts in bone marrow
* Peripheral blood white blood cell (WBC) count < 13,000/μL
* sEPO levels ≤ 500 mU/mL
* Non-transfusion dependence (NTD) according to IWG 2018 criteria
* Symptomatic anemia
* Age > 18 years
* Written informed consent

Exclusion Criteria:

* Patient does not accept bone marrow sampling during screening and during treatment
* Patient does not accept regular peripheral blood sampling for screening and during treatment.
* Patient does not accept subcutaneous application of LUS every three weeks
* Prior treatment for anemia associated with MDS (i.e. ESA, luspatercept), except previously treated with G-CSF/granulocyte-macrophage colony-stimulating factor (GM-CSF), both agents must be discontinued at least 4 weeks before registration
* Secondary MDS, i.e. MDS arising as the result of chemical injury or treatment with chemotherapy and/or radiation for other diseases
* Known clinically significant anemia due to iron, vitamin B12, or folate deficiencies, or autoimmune or hereditary hemolytic anemia, or gastrointestinal bleeding.
* Prior allogeneic or autologous stem cell transplant
* Prior history of AML
* Prior history of malignancies, other than MDS, unless the subject is free of the disease (including completion of any active or adjuvant treatment for prior malignancy) for ≥ 5 years.
* Major surgery within 8 weeks prior to registration.
* Uncontrolled hypertension, defined as repeated elevations of systolic blood pressure ≥160 mmHg or of diastolic blood pressure (DBP) ≥ 100 mmHg despite adequate treatment
* Platelet count < 30,000/μL (30 × 10^9/L)
* Estimated glomerular filtration rate or creatinine clearance < 40 mL/min
* Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) ≥ 3.0 × upper limit of normal (ULN)
* Alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) ≥ 3.0 × ULN
* Total bilirubin ≥ 2.0 × ULN
* Eastern Cooperative Oncology Group (ECOG) performance status > 2
* Stroke, deep venous thrombosis, pulmonary or arterial embolism within 6 months prior to registration
* Myocardial infarction, uncontrolled angina, uncontrolled heart failure, or uncontrolled cardiac arrhythmia within 6 months prior to registration.
* Subjects with a known ejection fraction of ˂ 35%, confirmed by a local echocardiography or multigated acquisition scan (MUGA) performed within 6 months prior to registration, are excluded
* Uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment), known human immunodeficiency virus (HIV), known evidence of active infectious hepatitis B, and/or known evidence of active hepatitis C.
* History of severe allergic or anaphylactic reactions or hypersensitivity to recombinant proteins or excipients in the IMP
* Subject has any significant medical condition, laboratory abnormality, psychiatric illness, or is considered vulnerable by local regulations (e.g., imprisoned or institutionalized) that would prevent the subject from participating in the study.
* Subject has any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she participates in the study
* Subject has any condition or concomitant medication that confounds the ability to interpret data from the study.
* Use of any of the following within five weeks prior to registration are prohibited: Anticancer cytotoxic chemotherapeutic agent or treatment, Corticosteroid, except for subjects on a stable or decreasing dose for ≥ 1 week prior to inclusion for medical conditions other than MDS, Iron chelation therapy, except for subjects on a stable or decreasing dose for at least 8 weeks prior to registration, Other RBC hematopoietic growth factors (e.g. interleukin [IL]-3)
* Pregnant or breastfeeding females
* Positive pregnancy test in women of childbearing potential.
* Female subjects of childbearing potential unwilling to use a highly effective method of contraception for the course of the study through 90 days after the last dose of study medication.
* Male subjects with procreative capacity not willing to use a highly effective method of contraception, starting with the first dose of study therapy through 90 days after the last dose of study therapy.
* Participation in other interventional trials.
* Patients under legal supervision or guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Estimated)
Dates: Start 2022-09-27 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Erythroid response (HI-E) | At the end of cycle 8 (each cycle is 21 days)
  To evaluate the proportion of patients who have an erythroid response (HI-E) according to the modified IWG 2018 criteria separately for four different clinical situations (cohorts) distinguished by two factors: Serum erythropoietin (sEPO) level AND Ring sideroblast (RS) status

SECONDARY OUTCOMES:
HI-E response (erythroid response) duration | From the date of treatment start until date of documented loss of response, assessed up to 18 months.]
  To evaluate HI-E response from the first day of response until loss of response.
Time to HI-E (erythroid response) | From the date of treatment start until first day of response, assessed up to end of cycle 8 (each cycle is 21 days)
  To evaluate the time between start of treatment and first day of response.
Neutrophil (HI-N) responses | At the end of cycle 8 (each cycle is 21 days)
  Neutrophil (HI-N) responses according to IWG 2018 criteria
Platelet (HI-P) responses | At the end of cycle 8 (each cycle is 21 days)
  Platelet (HI-P) responses according to IWG 2018 criteria
Safety of luspatercept (toxicities and adverse events) | From the date of treatment start until the end of study, assessed up to 48 months
  Assessments will include characterization of toxicities; characterization of AEs including type, incidence, severity, seriousness, and relationship to treatment
Impact of treatment assessed by using the validated European Organisation for Research and Treatment of Cancer Core Quality of Life questionnaire (EORTC QLQ-C30) | From the date of treatment start until the end of study, assessed up to 48 months.
  To assess patient-reported quality of life during luspatercept treatment: 30 questions assessing the quality of life of oncology patients across 10 subscales will be analyzed. All subscales have a score range from 0 to 100 points.
  Function subscales: a higher score represents a higher quality of life. Symptoms subscales: higher score represents higher level of symptoms/problems, i.e., represents lower quality of life.
Impact of luspatercept on quality of life by using the validated Quality of Life in Myelodysplasia Scale (QUALMS) | From the date of treatment start until the end of study, assessed up to 48 months
  QoL assessment using the QUALMS questionnaire up to end of treatment:
  38-item assessment tool for patients with Myelodysplastic Syndromes (MDS) QUALMS scores ranged from 24 to 99, with higher scores for better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Anne Sophie Kubasch, Dr., Principal Investigator — University Leipzig
Locations (22):
- Germany (22):
  - Praxis für Hämatologie und Onkologie Berlin-Mitte, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Carl-Thiem-Klinikum Cottbus gGmbH, Cottbus
  - OncoSearch Institut für klinische Studien GbR, Erlangen
  - Universitätsmedizin Greifswald Klinik Innere Medizin C / Hämatologie und Onkologie, Greifswald
  - OncoResearch Lerchenfeld GmbH, Hamburg
  - Klinikum Kassel GmbH Klinik für Hämatologie, Onkologie und Immunologie, Kassel
  - InVO Institut für Versorgungsforschung in der Onkologie GbR, Koblenz
  - VK&K Studien GbR, Landshut
  - Universität Leipzig - Medizinische Fakultät Klinik und Poliklinik für Hämatologie, Zelltherapie und Hämostaseologie, Leipzig
  - Mannheimer Onkologie Praxis, Mannheim
  - Universitätsklinikum Mannheim, III Medizinische Klinik - Hämatologie und Internistische Onkologie, Mannheim
  - Klinikum Hochsauerland GmbH, Meschede
  - Kliniken Maria Hilf GmbH Klinik für Hämatologie, Onkologie und Gastroenterologie, Mönchengladbach
  - Gemeinschaftspraxis Häamto-Onkologie, München
  - Klinikum rechts der Isar der TU München III. Medizinische Klinik - Hämatologie und Onkologie, München
  - Universitätsklinikum Münster, Medizinische Klinik A, Münster
  - Studiengesellschaft Onkologie Rhein/RuhrPraxis für Hämatologie und Onkologie Oberhausen und Düsseldorf, Oberhausen
  - Universitätsmedizin Rostock Klinik III (Hämatologie, Onkologie, Palliativmedizin) Zentrum für Innere Medizin, Rostock
  - Praxis ONKOSAAR Praxis für Hämatologie und Onkologie, Saarbrücken
  - Klinikum Mutterhaus, Trier
  - Universitätsklinikum Tübingen Medizinische Klinik II, AML/ALL/MDS, Tübingen

IPD SHARING:
Plan to Share IPD: No